CLINICAL TRIAL: NCT03320512
Title: P3 (Prepared, Protected, emPowered): Promoting Pre-exposure Prophylaxis (PrEP) Adherence Through a Social Networking, Gamification, and Adherence Support App
Brief Title: P3 (Prepared, Protected, emPowered)
Acronym: P3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Emory University (Other); Duke University (Other); Children's Hospital of Philadelphia (Other); The Fenway Institute (Other); Montefiore Medical Center (Other); Baylor College of Medicine (Other); Ruth M. Rothstein CORE Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 17-1951; 5U19HD089881-02 (NIH)
Record Dates: First submitted 2017-10-03; First posted 2017-10-25 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-08

CONDITIONS: Sexually Transmitted Diseases; Safe Sex; Adherence, Medication
Keywords: PrEP; gamification; mHealth; HIV prevention; truvada; eHealth; app; adherence; ymsm; transgender women
MeSH Terms: conditions — Sexually Transmitted Diseases; Safe Sex; Medication Adherence; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The trial will consist of a three-arm RCT to test intervention efficacy among young men who have sex with men (YMSM) and young transgender women who have sex with men (YTWSM) who are starting PrEP or are non-adherent to PrEP. Study arms will include P3, P3+, and standard of care (SOC). Participants will be recruited from seven cities. The investigators will enroll up to 240 participants and randomize them 1:1:1 to receive P3, P3+, or SOC. Assessments will be completed at months 0, 3, and 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- P3 (Experimental): Participants will use P3
  Interventions: Behavioral: P3
- P3+ (Experimental): Participants will use P3+
  Interventions: Behavioral: P3+
- Control (Placebo Comparator): Participants will receive the standard of care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: P3 — P3 is an interactive smartphone app that utilizes social networking and game-based mechanics to improve PrEP adherence and persistence in PrEP care. The participant will install P3 on their phone, receive a guided tour of the app and a reminder card with the research coordinator's phone number and email address and instructed to contact the research coordinator immediately to report difficulties with any app components or to report any problems with their phone or phone service. A help link is embedded within the app that directly links to study staff if assistance is needed. P3 arm participants will have 24-hour access to all features of P3.
  Other Names: Prepared, Protected, emPowered
  Arms: P3
Behavioral: P3+ — In P3+, participants receive all of P3 and the ability to text in the app with an adherence counselor, using Next Step Counseling (NSC). NSC is an interactive, client-centered motivational intervention to improve PrEP adherence. Key components of NSC include: review experiences with adherence, exploration of adherence facilitators and barriers, identification of adherence needs, identification of strategies to meet needs, and development of an adherence action plan. Participants will install P3+ on their phone. The adherence counselor feature will be unlocked for those in the P3+ arm. P3+ participants will have 24-hour access to all features of P3+.
  Arms: P3+
Behavioral: Control — Control participants will receive the standard of care for receiving a prescription for PrEP.
  Arms: Control

SUMMARY:
P3 (Prepared, Protected, emPowered) is an interactive smartphone app for HIV-uninfected YMSM and YTW that utilizes social networking and game-based mechanics as well as a comprehensive understanding of what constitutes "best practices" in app development to improve PrEP adherence and persistence in PrEP care.

DETAILED DESCRIPTION:
Sustainable, integrated PrEP adherence interventions are critically needed to reduce HIV incidence among YMSM and YTW. It is imperative that the investigators develop adherence interventions for YMSM and YTW initiating PrEP that are engaging, age-appropriate and take advantage of technologies that are already embedded in these individual's lives. A smartphone-delivered PrEP adherence intervention is well suited for this population, given they have a high-uptake and utilization of smartphone technology. The use of smartphones to deliver HIV prevention and care interventions has grown substantially in recent years due to: a) wide-scale adoption of smartphone technology among high-risk groups, b) the ability to deliver interventions in real-time within risk contexts, and c) low implementation costs.The accessibility, affordability, anonymity and acceptability of smartphones make them the intervention medium of choice for engaging youth and a logical platform to deliver an adherence intervention targeting PrEP. Further, smartphone interventions address can overcome issues that impede engagement with in-person interventions such as transportation logistics, stigma and confidentiality. Further youth, including YMSM and YTW are receptive to smartphone delivered interventions and these interventions can impact HIV related prevention behaviors.

P3 (Prepared, Protected, emPowered) is an interactive smartphone app for HIV-uninfected YMSM and YTW that utilizes social networking and game-based mechanics as well as a comprehensive understanding of what constitutes "best practices" in app development to improve PrEP adherence and persistence in PrEP care. Built on a successful, evidence-based platform designed and tested by our collaborating technology partner, Ayogo, P3 is flexible and responsive to changes in technology. This flexibility will also allow us to quickly respond to and modify our intervention to align with emerging PrEP practice standards and guidelines.

Despite the benefits of app-based interventions, maintaining engagement over time can be particularly challenging. Lack of rapport building may contribute to lower retention rates in technology-based interventions. Further, the available literature suggests that some tools, including technology based tools, may be more beneficial to patient adherence when combined with education or counseling. To investigate this possibility, the investigators will include a study arm (P3+) that includes P3 and adherence counseling delivered by a counselor through the P3 app.

This study has three phases, usability testing, field testing, and a randomized-controlled trial (RCT). In usability testing the investigators will test beta versions of the app and gain feedback about the intervention from the target population, identify any technical issues, and get feedback on app content. Field testing is to ensure that the features, platform and content of P3 and P3+ are acceptable to the target population and that there are no technical challenges or user concerns with either the app, the dried blood spot (DBS), hair, or mitra sampling collection.

The last phase is a three arm, RCT that will test the efficacy of P3, a novel, theory-based mobile app that utilizes game mechanics and social networking features to improve PrEP adherence, retention in PrEP clinical care, and PrEP persistence among young men who have sex with men (YMSM) and young trans women (YTW) who have sex with men, ages 16-24. The investigators will test the efficacy of P3 and P3+, which adds Next Step Counseling delivered by an adherence counselor through the app, against PrEP standard of care. Participants will be randomized to P3, P3+, or standard of care. A cost comparison between P3 and P3+ will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 16-24
* Were assigned male sex at birth
* Report sex with men or transgender women
* Are able to speak and read English
* Have reliable daily access to an Android or iOS smartphone with a data plan
* Are HIV-uninfected (self-report)
* Are not currently on PrEP but plan to initiate in the next 7 days and have an active PrEP prescription (prescription confirmed by study staff) OR on PrEP have an active PrEP prescription (prescription confirmed by study staff)
* Recruited from one of 9 subject recruitment venues (SRV) cities (Atlanta, Georgia; Boston, Massachusetts; Bronx, New York; Chicago, Illinois; Houston, Texas; Philadelphia, Pennsylvania; Tampa, Florida; Chapel Hill, NC; Charlotte, NC)

Exclusion Criteria:

* Aged younger than 15 years or older than 24 years
* Not available to meet with project staff for planned study visit(s)
* Non-English speaking
* Living with HIV
* Not currently prescribed PrEP (study staff unable to verify participant has an active PrEP prescription by a health provider)
* Anticipate not having reliable access to a smartphone with a data plan for 2 or more days during field testing or 1 or more weeks during the RCT intervention period
* Planning to move out of study area during the study period
* Unwilling or unable to comply with protocol requirements.
* Participated in field trial phase of P3 study
* Unable to be consented due to active substance use or psychological condition.

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self-identify as MSM or TW who has sex with men
Enrollment: 246 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Weidman, MD, Principal Investigator — UNC Chapel Hill
Locations (9):
- United States (9):
  - University of South Florida Infectious Diseases, Tampa, Florida
  - PRISM Health, Atlanta, Georgia
  - The Adolescent and Young Adult Research (AYAR) at the CORE Center, Chicago, Illinois
  - The Fenway Institute, Boston, Massachusetts
  - Children's Hospital at Montefiore, The Bronx, New York
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - RAIN, Charlotte, North Carolina
  - Adolescent Initiative at Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams MP, Manjourides J, Smith LH, Rainer CB, Hightow-Weidman LB, Haley DF. Studying the Digital Intervention Engagement-Mediated Relationship Between Intrapersonal Measures and Pre-Exposure Prophylaxis Adherence in Sexual and Gender Minority Youth: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2025 Jan 13;27:e57619. doi: 10.2196/57619. PMID 39804696
- [Derived] Yigit I, Budhwani H, Rainer CB, Claude K, Muessig KE, Hightow-Weidman LB. Associations Between PrEP Stigma, PrEP Confidence, and PrEP Adherence: Conditional Indirect Effects of Anticipated HIV Stigma. J Acquir Immune Defic Syndr. 2024 Oct 1;97(2):99-106. doi: 10.1097/QAI.0000000000003474. PMID 39250643
- [Derived] Budhwani H, Yigit I, Maragh-Bass AC, Rainer CB, Claude K, Muessig KE, Hightow-Weidman LB. Validation of HIV Pre-Exposure Prophylaxis (PrEP) Medication Scales with Youth on PrEP: PrEP Confidence Scale and PrEP Difficulties Scale. AIDS Patient Care STDS. 2022 Nov;36(11):443-450. doi: 10.1089/apc.2022.0072. Epub 2022 Oct 27. PMID 36306520
- [Derived] LeGrand S, Knudtson K, Benkeser D, Muessig K, Mcgee A, Sullivan PS, Hightow-Weidman L. Testing the Efficacy of a Social Networking Gamification App to Improve Pre-Exposure Prophylaxis Adherence (P3: Prepared, Protected, emPowered): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Dec 18;7(12):e10448. doi: 10.2196/10448. PMID 30563818

RESULTS

PARTICIPANT FLOW:
Groups:
- P3 Application: Participants will use P3
  P3: P3 is an interactive smartphone app that utilizes social networking and game-based mechanics to improve PrEP adherence and persistence in Pre-Exposure Prophylaxis (PrEP) care. The participant will install P3 on their phone, receive a guided tour of the app and a reminder card with the research coordinator's phone number and email address and instructed to contact the research coordinator immediately to report difficulties with any app components or to report any problems with their phone or phone service. A help link is embedded within the app that directly links to study staff if assistance is needed. P3 arm participants will have 24-hour access to all features of P3.
- P3+ Application: Participants will use P3+
  P3+: In P3+, participants receive all of P3 and the ability to text in the app with an adherence counselor, using Next Step Counseling (NSC). NSC is an interactive, client-centered motivational intervention to improve PrEP adherence. Key components of NSC include: review experiences with adherence, exploration of adherence facilitators and barriers, identification of adherence needs, identification of strategies to meet needs, and development of an adherence action plan. Participants will install P3+ on their phone. The adherence counselor feature will be unlocked for those in the P3+ arm. P3+ participants will have 24-hour access to all features of P3+.
Period: Overall Study
Arm/Group | P3 Application | P3+ Application | Control
Started | 82 | 81 | 83
Month 3 Survey Started | 69 | 72 | 71
Month 3 Survey Completed | 69 | 72 | 68
Month 3 Lab Sample Collected | 51 | 54 | 51
Month 6 Survey Started | 67 | 72 | 69
Month 6 Survey Completed | 65 | 71 | 68
Month 6 Lab Sample Collected | 53 | 59 | 51
Completed | 82 | 81 | 83
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- P3 Application: Participants will use P3
  P3: P3 is an interactive smartphone app that utilizes social networking and game-based mechanics to improve PrEP adherence and persistence in PrEP care. The participant will install P3 on their phone, receive a guided tour of the app and a reminder card with the research coordinator's phone number and email address and instructed to contact the research coordinator immediately to report difficulties with any app components or to report any problems with their phone or phone service. A help link is embedded within the app that directly links to study staff if assistance is needed. P3 arm participants will have 24-hour access to all features of P3.
- Total: Total of all reporting groups
Arm/Group | P3 Application | P3+ Application | Control | Total
Number analyzed (Participants) | 82 | 81 | 83 | 246
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [20 to 23] | 22 [20 to 23] | 22 [21 to 23] | 22 [20 to 23]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 71 | 71 | 74 | 216
  Trans female, trans woman, or transfeminine | 0 | 3 | 2 | 5
  Genderqueer, gender non-conforming, or non-binary | 3 | 2 | 4 | 9
  Multiple genders reported | 8 | 3 | 3 | 14
  Declined to answer | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 82 | 81 | 83 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 18 | 27 | 71
  Not Hispanic or Latino | 56 | 63 | 56 | 175
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 7 | 5 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 19 | 16 | 51
  White | 49 | 46 | 42 | 137
  More than one race | 3 | 4 | 9 | 16
  Unknown or Not Reported | 6 | 6 | 11 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82 | 81 | 83 | 246

OUTCOME MEASURES:

1. Primary Outcome: PrEP Adherence Defined by Tenofovir Diphosphate (P3 and P3+ vs Control)
Description: PrEP adherence is measured by blood sample levels of tenofovir diphosphate (TFV-DP) with blood concentration consistent with > 4 doses/week at 3- and 6- month follow-ups. The estimation of the average treatment effect compared P3 and P3+ combined to Control.
Time Frame: Month 3, Month 6
Population: Data were included if 3- and/or 6-month samples were available. A participant's data was available if at least one sample was returned and that sample was readable (i.e., sample was not degraded and participant was not using Descovy).
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 38 | 52 | 45
Participants
  Month 3: number analyzed (Participants) | 32 | 41 | 35
  Month 3 | 24 | 33 | 23
  Month 6: number analyzed (Participants) | 29 | 42 | 34
  Month 6 | 18 | 25 | 20
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population; Test type: Superiority; p = 0.04965, TMLE estimation of ATE and Wald test; Targeted Maximum Likelihood Estimation (TMLE) Average Treatment Effect (ATE); Average Treatment Effect = 0.15, 95% CI 2-sided [0.00 to 0.29]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population; Test type: Superiority; p = 0.62, TMLE estimation of ATE and Wald test; Average Treatment Effect = -0.04, 95% CI 2-sided [-0.21 to 0.13]

2. Primary Outcome: PrEP Adherence Defined by Emtricitabine Triphosphate (P3 and P3+ vs Control)
Description: PrEP adherence is measured by blood sample levels of emtricitabine triphosphate (FTC-TP) with blood concentration consistent with > 4 doses/week at 3- and 6- month follow-ups. The estimation of the average treatment effect compared P3 and P3+ combined to Control.
Time Frame: Month 3, Month 6
Population: Data were included if 3- and/or 6-month samples were available. A participant's data was available if at least one sample was returned and that sample was readable (i.e., sample was not degraded).
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 62 | 69 | 64
Participants
  Month 3: number analyzed (Participants) | 50 | 54 | 51
  Month 3 | 36 | 38 | 29
  Month 6: number analyzed (Participants) | 50 | 56 | 48
  Month 6 | 31 | 31 | 24
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population; Test type: Superiority; p = 0.11, TMLE estimation of ATE and Wald test; Average Treatment Effect = 0.12, 95% CI 2-sided [-0.03 to 0.26]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population; Test type: Superiority; p = 0.38, TMLE estimation of ATE and Wald test; Average Treatment Effect = 0.06, 95% CI 2-sided [-0.08 to 0.21]

3. Secondary Outcome: Number of Participants With Self-reported Retention in PrEP Clinical Care
Description: The investigators define "retention in care" as at least 1 PrEP clinical visit occurring in the last 3 months.
Time Frame: Month 3, Month 6
Population: Data were included if 3- and/or 6-month samples were available. A participant's data was available if they sufficiently responded to the clinical care survey questions and the survey was submitted within appropriate time window.
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 73 | 75 | 74
Participants
  Month 3: number analyzed (Participants) | 66 | 70 | 69
  Month 3 | 38 | 43 | 38
  Month 6: number analyzed (Participants) | 64 | 70 | 68
  Month 6 | 32 | 34 | 25
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.68, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = 0.04, 95% CI 2-sided [-0.09 to 0.16]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.53, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = 0.11, 95% CI 2-sided [-0.03 to 0.25]

4. Secondary Outcome: PrEP Persistence
Description: PrEP persistence will be measured by self-report at follow up of current PrEP use.
Time Frame: Month 3, Month 6
Population: Data were included if 3- and/or 6-month responses were available. A participant's data was available if they sufficiently responded to the PrEP persistence survey questions and the survey was submitted within appropriate time window.
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 74 | 77 | 74
Participants
  Month 3: number analyzed (Participants) | 69 | 71 | 69
  Month 3 | 66 | 64 | 59
  Month 6: number analyzed (Participants) | 66 | 71 | 69
  Month 6 | 52 | 49 | 52
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.53, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = 0.06, 95% CI 2-sided [-0.02 to 0.15]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.96, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = 0, 95% CI 2-sided [-0.12 to 0.12]

5. Secondary Outcome: Insertive Condomless Anal Sex
Description: Sexual Practices were assessed by self-reported number of insertive condomless anal sex occurrences during the past 3 months. This question is asked at the 3- and 6-month follow-up surveys.
Time Frame: Month 3, Month 6
Population: Data were included if 3- and/or 6-month responses were available. A participant's data was available if they sufficiently responded to the sexual activity survey questions and the survey was submitted within appropriate time window.
Measure: Median (Inter-Quartile Range); unit: sex acts
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 73 | 77 | 73
sex acts
  Month 3: number analyzed (Participants) | 69 | 72 | 69
  Month 3 | 1 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
  Month 6: number analyzed (Participants) | 65 | 72 | 69
  Month 6 | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.93, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = 0.08, 95% CI 2-sided [-0.84 to 1.00]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.60, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -1.12, 95% CI 2-sided [-4.16 to 1.91]

6. Secondary Outcome: Receptive Condomless Anal Sex
Description: Sexual Practices were assessed by self-reported number of receptive condomless anal sex occurrences during the past 3 months. This question is asked at the 3- and 6-month follow-up surveys.
Time Frame: Month 3, Month 6
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: sex acts
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 73 | 77 | 73
sex acts
  Month 3: number analyzed (Participants) | 69 | 72 | 69
  Month 3 | 1 [0 to 3] | 0 [0 to 2] | 1 [0 to 3]
  Month 6: number analyzed (Participants) | 65 | 72 | 69
  Month 6 | 1 [0 to 3] | 0 [0 to 1] | 0 [0 to 2]
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.60, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = 0.73, 95% CI 2-sided [-1.03 to 2.48]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.60, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -0.91, 95% CI 2-sided [-2.86 to 1.04]

7. Secondary Outcome: Sexually Transmitted Infections (STI) Incidence
Description: Self-reported STIs (combined rectal and urethral gonorrhea and chlamydia, syphilis) in last 3 months. This question is asked at the 3- and 6-month follow-up surveys.
Time Frame: Month 3, Month 6
Population: Data were included if 3- and/or 6-month responses were available. A participant's data was available if they sufficiently responded to the STI survey questions and the survey was submitted within appropriate time window.
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 54 | 60 | 55
Participants
  Month 3 Gonorrhea: number analyzed (Participants) | 43 | 51 | 41
  Month 3 Gonorrhea | 12 | 14 | 14
  Month 6 Gonorrhea: number analyzed (Participants) | 37 | 40 | 38
  Month 6 Gonorrhea | 11 | 6 | 10
  Month 3 Chlamydia: number analyzed (Participants) | 43 | 51 | 41
  Month 3 Chlamydia | 11 | 14 | 17
  Month 6 Chlamydia: number analyzed (Participants) | 37 | 40 | 38
  Month 6 Chlamydia | 11 | 8 | 12
  Month 3 Syphilis: number analyzed (Participants) | 43 | 51 | 41
  Month 3 Syphilis | 9 | 8 | 12
  Month 6 Syphilis: number analyzed (Participants) | 37 | 40 | 38
  Month 6 Syphilis | 11 | 3 | 9
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 Gonorrhea The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.60, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -0.06, 95% CI 2-sided [-0.20 to 0.08]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 Gonorrhea The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.60, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -0.06, 95% CI 2-sided [-0.21 to 0.09]
Statistical Analysis 3: Comparison: P3 Application vs P3+ Application vs Control; Month 3 Chlamydia The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.53, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -0.13, 95% CI 2-sided [-0.30 to 0.03]
Statistical Analysis 4: Comparison: P3 Application vs P3+ Application vs Control; Month 6 Chlamydia The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.60, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -0.08, 95% CI 2-sided [-0.24 to 0.08]
Statistical Analysis 5: Comparison: P3 Application vs P3+ Application vs Control; Month 3 Syphillis The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.53, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -0.11, 95% CI 2-sided [-0.25 to 0.04]
Statistical Analysis 6: Comparison: P3 Application vs P3+ Application vs Control; Month 6 Syphillis The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.60, TMLE estimation of ATE and Wald test — P-values adjusted using the Benjamini Hochberg procedure; Average Treatment Effect = -0.07, 95% CI 2-sided [-0.20 to 0.07]

8. Secondary Outcome: PrEP Adherence Defined by Tenofovir Diphosphate (P3 vs Control and P3+ vs Control)
Description: PrEP adherence is measured by blood sample levels of tenofovir diphosphate (TFV-DP) with blood concentration consistent with > 4 doses/week at 3- and 6- month follow-ups. The estimation of the average treatment effect compared P3 to Control and also P3+ to Control.
Time Frame: Month 3, Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 38 | 52 | 45
Participants
  Month 3: number analyzed (Participants) | 32 | 41 | 35
  Month 3 | 24 | 33 | 23
  Month 6: number analyzed (Participants) | 29 | 42 | 34
  Month 6 | 18 | 25 | 20
Statistical Analysis 1: Comparison: P3 Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 vs. Control; Test type: Superiority; Average Treatment Effect = 0.11, 95% CI 2-sided [-0.07 to 0.29] — TMLE estimation of ATE and Wald Confidence Interval
Statistical Analysis 2: Comparison: P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3+ vs. Control; Test type: Superiority; Average Treatment Effect = 0.19, 95% CI 2-sided [0.03 to 0.34] — TMLE estimation of ATE and Wald Confidence Interval
Statistical Analysis 3: Comparison: P3 Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 vs. Control; Test type: Superiority; Average Treatment Effect = -0.06, 95% CI 2-sided [-0.27 to 0.15] — TMLE estimation of ATE and Wald Confidence Interval
Statistical Analysis 4: Comparison: P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3+ vs. Control; Test type: Superiority; Average Treatment Effect = -0.02, 95% CI 2-sided [-0.21 to 0.16] — TMLE estimation of ATE and Wald Confidence Interval

9. Secondary Outcome: PrEP Adherence Defined by Emtricitabine Triphosphate (P3 vs Control and P3+ vs Control)
Description: PrEP adherence is measured by blood sample levels of emtricitabine triphosphate (FTC-TP) with blood concentration consistent with > 4 doses/week at 3- and 6- month follow-ups. The estimation of the average treatment effect compared P3 to Control and also P3+ to Control.
Time Frame: Month 3, Month 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 62 | 69 | 64
Participants
  Month 3: number analyzed (Participants) | 50 | 54 | 51
  Month 3 | 36 | 38 | 29
  Month 6: number analyzed (Participants) | 50 | 56 | 48
  Month 6 | 31 | 31 | 24
Statistical Analysis 1: Comparison: P3 Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 vs. Control; Test type: Superiority; Average Treatment Effect = 0.11, 95% CI 2-sided [-0.05 to 0.26] — TMLE estimation of ATE and Wald Confidence Interval
Statistical Analysis 2: Comparison: P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3+ vs. Control; Test type: Superiority; Average Treatment Effect = 0.13, 95% CI 2-sided [-0.04 to 0.29] — TMLE estimation of ATE and Wald Confidence Interval
Statistical Analysis 3: Comparison: P3 Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 vs. Control; Test type: Superiority; Average Treatment Effect = 0.09, 95% CI 2-sided [-0.08 to 0.26] — TMLE estimation of ATE and Wald Confidence Interval
Statistical Analysis 4: Comparison: P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3+ vs. Control; Test type: Superiority; Average Treatment Effect = 0.03, 95% CI 2-sided [-0.13 to 0.19] — TMLE estimation of ATE and Wald Confidence Interval

10. Secondary Outcome: Self-Reported Weekly PrEP Use
Description: Number of participants reported taking their PrEP medication >/= 4 days in the past week.
Time Frame: Month 3, Month 6
Population: Data were included if 3- and/or 6-month responses were available. A participant's data was available if they sufficiently responded to the PrEP use survey questions and the survey was submitted within appropriate time window.
Measure: Count of Participants; unit: Participants
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 73 | 77 | 74
Participants
  Month 3: number analyzed (Participants) | 65 | 63 | 59
  Month 3 | 58 | 59 | 51
  Month 6: number analyzed (Participants) | 52 | 49 | 51
  Month 6 | 49 | 48 | 47
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.11, TMLE estimation of ATE and Wald test; Average Treatment Effect = 0.09, 95% CI 2-sided [-0.02 to 0.19]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.82, TMLE estimation of ATE and Wald test; Average Treatment Effect = -0.01, 95% CI 2-sided [-0.14 to 0.11]

11. Secondary Outcome: Self-Reported Monthly PrEP Use
Description: Median self-reported percent of time in the past month that participants' took their PrEP as prescribed.
Time Frame: Month 3, Month 6
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: percentage of time compliant
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 74 | 77 | 74
percentage of time compliant
  Month 3: number analyzed (Participants) | 69 | 70 | 70
  Month 3 | 100 [80 to 100] | 100 [90 to 100] | 90 [72.5 to 100]
  Month 6: number analyzed (Participants) | 66 | 71 | 68
  Month 6 | 90 [50 to 100] | 90 [25 to 100] | 90 [67.5 to 100]
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application vs Control; Month 3 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.05, TMLE estimation of ATE and Wald test — The a priori threshold for statistical significance is 0.025; Average Treatment Effect = 8.95, 95% CI 2-sided [0.07 to 17.83]
Statistical Analysis 2: Comparison: P3 Application vs P3+ Application vs Control; Month 6 The analysis includes the intent-to-treat population and compares P3 and P3+ vs. Control; Test type: Superiority; p = 0.45, TMLE estimation of ATE and Wald test; Average Treatment Effect = -3.69, 95% CI 2-sided [-13.33 to 5.95]

12. Secondary Outcome: Mean Site-Level Intervention Cost
Description: Information was collected on (1) time spent by study staff for training and supervision of adherence counselor(s); (2) time participants spent in the adherence counseling sessions; and (3) costs associated with the delivery of both P3 and P3+. Resources were organized into standard expenditure categories and attributed to the corresponding P3 or P3+ arm and study site as appropriate.
Time Frame: Throughout the duration of the study, approximately 1.5 years
Population: This outcome pertains to participating sites rather than actual participants. The analysis was applicable only to the intervention arms; the control arm is excluded since there was no intervention or associated cost. Data were not reported for 1 site which was inactive during the data collection periods.
Measure: Mean (Standard Deviation); unit: average cost per participant in USD
Units Other Than Participants: Participating Sites
Arm/Group | P3 Application | P3+ Application | Control
Number analyzed (Participants) | 32 | 41 | 0
Number analyzed (Participating Sites) | 8 | 8 | 0
average cost per participant in USD | 551.88 (160.43) | 673.52 (161.06) |
Statistical Analysis 1: Comparison: P3 Application vs P3+ Application; Participants were included if they were at an active site with cost data and had a 3-month binary TFV measure; Test type: Superiority; Incremental cost effectiveness ratio = 25.79, 95% CI 2-sided [-194.05 to 236.81] — The confidence interval was created using percentile bootstrap

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of the Informed consent by each participant until the end of the study, a duration of up to 6 months.
Arm/Group | P3 Application | P3+ Application | Control
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/81 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81 | 0/83
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81 | 0/83

LIMITATIONS AND CAVEATS:
Despite the sample including about a quarter Black (20.7%) and another quarter Hispanic or Latinx (28.9%) participants, a majority of the sample was White (55.7%). And while the study was conducted across nine U.S. cities (Atlanta, Boston, Chicago, Chapel Hill, Charlotte, Houston, New York, Philadelphia, and Tampa) the results may not be generalizable to entire populations of young men who have sex with men (YMSM) and young transgender women who have sex with men (YTWSM).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03320512/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03320512/SAP_001.pdf